CLINICAL TRIAL: NCT03413020
Title: Efficacy of Tailored for Helicobacter Pylori Rescue Treatment Based on Antimicrobial-susceptibility Testing
Brief Title: Tailored Therapy for Helicobacter Pylori Rescue Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Hong Lu, MD, Medical Doctor of Division of Gastroenterology and Hepatology of Renji Hospital,Professor of Medicine, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: rjkls2017198
Record Dates: First submitted 2018-01-22; First posted 2018-01-29 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; Rescue therapy; Tailored therapy; Antimicrobial susceptibility testing
MeSH Terms: interventions — Esomeprazole; Amoxicillin; Clarithromycin; Metronidazole; Levofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tailored Therapy (Experimental): After antimicrobial susceptibility testing of Helicobacter pylori from biopsy samples, according to antibiotic resistance pattern of each one, give esomeprazole, amoxicillin and one sensitive of clarithromycin, metronidazole and levofloxacin.If isolates were resistant to all three tested antibiotics, give esomeprazole, bismuth potassium citrate, metronidazole and amoxicillin for 14 days.
  Interventions: Drug: esomeprazole; Drug: bismuth Potassium Citrate; Drug: amoxicillin; Drug: clarithromycin; Drug: metronidazole; Drug: levofloxacin

INTERVENTIONS:
Drug: esomeprazole — proton pump inhibitor
Drug: bismuth Potassium Citrate — gastric mucosal protective drug with anti-H. pylori effect
Drug: amoxicillin — antibiotic for H. pylori eradication
Drug: clarithromycin — antibiotic for H. pylori eradication
Drug: metronidazole — antibiotic for H. pylori eradication
Drug: levofloxacin — antibiotic for H. pylori eradication

SUMMARY:
With increasing antibiotic resistance and unsatisfactory results of empiric eradication regimens, tailored therapy may be the best choice to achieve high efficacy for rescue treatment. This study aimed to evaluate the eradication rates, safety, and compliance of antimicrobial susceptibility-based tailored therapy for rescue treatment in patients with Helicobacter pylori infection.

ELIGIBILITY:
Inclusion Criteria:

* Participants with non-ulcer functional dyspepsia or scarred peptic ulcer disease
* Previous failures of H. pylori eradication therapy and need rescue therapy
* Ability and willingness to participate in the study and to sign and give informed consent
* Confirmed H. pylori infection

Exclusion Criteria:

* Less than 18 years old
* With previous gastric surgery
* Major systemic diseases
* Pregnancy or lactation
* Allergy to any of the study drugs
* Administration of antibiotics, bismuth, antisecretory drugs in 8 weeks prior to inclusion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Helicobacter pylori eradication rate | Six weeks after completion of therapy
  Six weeks after completion of therapy, H. pylori eradication was assessed by ¹³C-urea breath test. Eradication was defined as negative result from urea breath test (<4‰) (4‰ as the cutoff value).

SECONDARY OUTCOMES:
Rate of adverse effects | Within 7 days after completion of therapy
  The subjects were asked to grade the severity of adverse events according to their influence on daily activities, experienced as "mild" (transient and well tolerated), "moderate" (causing discomfort and partially interfering with daily activities), or "severe" (causing considerable interference with daily activities).
Compliance rate | Within 7 days after completion of therapy
  Compliance was defined as poor when they had taken less than 80% of the total medication.

OTHER OUTCOMES:
Medical cost per patient of tailored therapy | Two months after completion of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Hong Lu, M.D., Principal Investigator — Renji Hospital, School of Medicine, Shanghai Jiao Tong University
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yu L, Luo L, Long X, Liang X, Ji Y, Chen Q, Song Y, Li X, Graham DY, Lu H. Susceptibility-guided therapy for Helicobacter pylori infection treatment failures. Therap Adv Gastroenterol. 2019 Sep 9;12:1756284819874922. doi: 10.1177/1756284819874922. eCollection 2019. PMID 31523279